CLINICAL TRIAL: NCT06794762
Title: Examination of the Effects of Core Stabilization Exercises on Physical Function, Functional Muscle Strength, Functional Exercise Capacity, Postural Control and Fatigue in Children with Acute Lymphoblastic Leukemia Receiving Maintenance Treatment
Brief Title: Effects of Core Stabilization Exercises in Children with Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Melike Müsevitoğlu, Melike Müsevitoğlu, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024/023-12
Record Dates: First submitted 2025-01-13; First posted 2025-01-27 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; Maintenance Chemotherapy; Rehabilitation; Exercise; Core Stabilization Exercises; Cancer; Physical Function; Functional Muscle Strength; Functional Exercise Capacity; Postural Control; Fatigue
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Motor Activity; Neoplasms; Fatigue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Experimental): Exercises will be applied to the participants participating in the study 3 days a week, 8 weeks, and 24 sessions in total.
  Interventions: Other: Conventional exercises
- Intervention group (Experimental): Exercises will be applied to the individuals participating in the study 3 days a week, 8 weeks, and 24 sessions in total. Exercises will be applied after the conventional therapy sessions.
  Interventions: Other: Core stabilization exercises in addition to conventional exercises

INTERVENTIONS:
Other: Conventional exercises — Aerobic exercise and stretching exercises will be applied in the conventional exercise program.
  A 20-30 minute walking will be done as aerobic exercise. Stretching exercises will be done for major muscle groups in 3 sets and 10 repetitions.
  Arms: Control group
Other: Core stabilization exercises in addition to conventional exercises — In addition to the conventional exercise program, core stabilization exercises will be applied. During the exercises, participants will be trained on neutralizing the spine and working the transverse abdominis and multifidus muscles, correct postural control, and performing the exercises with diaphragmatic breathing.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to investigate the effects of core stabilization exercises applied in addition to the conventional exercise program on physical function, functional muscle strength, functional exercise capacity, postural control and fatigue in children with acute lymphoblastic leukemia receiving maintenance treatment.

Participants will be divided into two groups; the first group will be given a conventional exercise program, while the second group will be given core stabilization exercises in addition to the conventional exercise program.

DETAILED DESCRIPTION:
Acute Lymphoblastic Leukemia (ALL) is a malignancy resulting from the abnormal proliferation of lymphoid cells that can invade the bone marrow, blood, and extramedullary regions, and it is the most common malignancy in childhood. Specific chemotherapy-related problems are frequently observed in children with ALL. These include a reduction in cardiopulmonary fitness, balance, posture, proximal muscle strength, and flexibility, as well as postural control issues and functional mobility impairments, in addition to fatigue.

The aim of this study is to investigate the effects of core stabilization exercises, applied in addition to a conventional exercise program, on physical function, functional muscle strength, functional exercise capacity, postural control, and fatigue in children with Acute Lymphoblastic Leukemia undergoing maintenance therapy.

Participants will be divided into two groups: the first group will follow a conventional exercise program, while the second group will receive core stabilization exercises in addition to the conventional program. All participants will be randomly assigned to the groups using the software available at http://www.randomizer.org. The exercise sessions will be conducted three times a week for a total of 8 weeks, with 24 sessions in total. Demographic information will be recorded for participants who agree to take part in the study and meet the inclusion criteria. The scales and tests designed to assess the participants' physical function, functional muscle strength, functional exercise capacity, postural control, and fatigue will be administered both before and after the study.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7-18
* Diagnosed with ALL
* In the maintenance phase of chemotherapy
* Children without acute thrombosis, active ischemia, hemodynamic instability
* Children without uncontrolled pain
* Children who can follow verbal instructions.

Exclusion Criteria:

* Children who have received or are receiving cranial radiotherapy
* Children with any cardiovascular disease, acute or chronic respiratory disease
* Children with acute or chronic bone, joint, muscle problems
* Children diagnosed with neuromotor deficits or genetic disorders
* Children with vision problems other than refractive errors

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go Test (TUG) | Before 8 weeks of treatment
  This test aims to evaluate the physical function.
Timed Up and Go Test (TUG) | After 8 weeks of treatment
  This test aims to evaluate the physical function.
Sit-up Test | Before 8 weeks of treatment
  This test aims to evaluate the functional muscle strength
Sit-up Test | After 8 weeks of treatment
  This aims to evaluate the functional muscle strength.
6-Minute Walk Test | Before 8 weeks of treatment
  This test aims to evaluate the functional exercise capacity.
6-Minute Walk Test | After 8 weeks of treatment
  This test aims to evaluate the functional exercise capacity.
Balance Error Scoring System | Before 8 weeks of treatment
  This test aims to evaluate the postural control.
Balance Error Scoring System | After 8 weeks of treatment
  This test aims to evaluate the postural control.
Pediatric Quality of Life Multidimensional Fatigue Scale | Before 8 weeks of treatment
  This scale aims to evaluate the fatigue in pediatric patients.
Pediatric Quality of Life Multidimensional Fatigue Scale | After 8 weeks of treatment
  This scale aims to evaluate the fatigue in pediatric patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No